CLINICAL TRIAL: NCT01118052
Title: A Phase II Evaluation of Intraperitoneal EGEN-001 (IL-12 Plasmid Formulated With PEG-PEI-Cholesterol Lipopolymer) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: EGEN-001 in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170Q; NCI-2011-02041 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FD-R-003942; CDR0000672159; GOG-0170Q (Other: NRG Oncology); GOG-0170Q (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-08

CONDITIONS: Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — GEN-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (EGEN-001) (Experimental): Patients receive intraperitoneal EGEN-001 on days 1, 8, 15, and 22. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: PEG-PEI-cholesterol Lipopolymer-encased IL-12 DNA Plasmid Vector GEN-1

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: PEG-PEI-cholesterol Lipopolymer-encased IL-12 DNA Plasmid Vector GEN-1 — Given intraperitoneally

SUMMARY:
This phase II trial studies the side effects and how well EGEN-001 works in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer that is persistent or has come back. Biological therapies, such as EGEN-001, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop tumor cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial) in patients with persistent or recurrent ovarian epithelial, fallopian tube, or primary peritoneal carcinoma.

II. To determine the frequency and severity of adverse events as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To collect blood and peritoneal lavage fluid from patients that will be stored for future research.

OUTLINE:

Patients receive intraperitoneal EGEN-001 on days 1, 8, 15, and 22. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI; patients must have evidence of intra-abdominal/pelvic disease; patients with disease exclusively located outside of the abdominal/pelvic cavity are not eligible
* Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2

  * Patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy:

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted therapy and immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment
* Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

  * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
  * Note: patients on this non-cytotoxic study are allowed to receive additional cytotoxic chemotherapy for management of recurrent or persistent disease, as defined above; however, due to the novel nature of biologic compounds, patients are encouraged to enroll on second-line non-cytotoxic studies prior to receiving additional cytotoxic therapy
* Absolute neutrophil count (ANC) greater or equal to 1,500/mcl
* Platelet count greater or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x upper limit of normal (ULN) OR calculated creatinine clearance greater than or equal to 50 mL/min; any evidence of renal obstruction must be corrected prior to treatment
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) aspartate aminotransferase (AST) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neuropathy (sensory or motor) less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have had previous treatment with EGEN-001
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted above are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with a past history of primary endometrial cancer are excluded unless all of the following conditions are met: stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients with a serious uncontrolled medical illness or disorder, abdominal surgery (for reasons other than IP port placement) or active infection within four weeks of study entry; patients may have surgery for the purpose of IP port placement greater than or equal to one week(s) before study entry and treatment
* Patients with any condition/anomaly that would interfere with the appropriate placement of the IP catheter for study drug administration including: abdominal surgery within 4 weeks of study entry (for reasons other than IP port placement), intestinal dysfunction or suspected extensive adhesions from prior history or finding at laparoscopy
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Alvarez, Principal Investigator — NRG Oncology
Locations (11):
- United States (11):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Case Western Reserve University, Cleveland, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG 170Q accrued 22 patients from November 2010 to January 2013.
Period: Overall Study
Arm/Group | Treatment (EGEN-001)
Started | 22
Completed | 20
Not Completed | 2
Not completed — Never treated | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (EGEN-001)
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 0
  40 - 49 years | 1
  50 - 59 years | 12
  60 - 69 years | 5
  70 - 79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Survive Progression-free for at Least 6 Months
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1. RECIST 1.1 defines progressive disease as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or unequivocal progression of non-target lesions is also considered progression
Time Frame: Every other cycle during treatment, then every 3 months until disese progression is confirmed, up to 5 years
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (EGEN-001)
Number analyzed (Participants) | 20
Participants
  Patients with Progression Free Survival > 6 months | 6
  Patients with Progression Free Survival < 6 months | 14

2. Primary Outcome: Patients Who Have Objective Tumor Response (Complete or Partial Response)
Description: Complete and Partial Tumor Response by RECIST 1.1. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: CT or MRI used to follow lesion for measurable disease every other cycle. Patient's best response while on study treatment was recorded, Up to 5 years
Population: Eligible and Treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (EGEN-001)
Number analyzed (Participants) | 20
percentage of participants | 0.0 [0.0 to 13.9]

3. Primary Outcome: Adverse Events Deemed at Least Possibly Related to Treatment, as Assessed by NCI CTCAE Version 4.0
Description: Adverse events are listed by adverse event and grade. The number of participants affected is listed.
Time Frame: All Adverse Events (AEs) deemed at least possibly related to study treatmetn occurring during treatment and up to 30 days after stopping the study treatment. for up to 5 years after stopping study treatment
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 4.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 4.0
- Grade 2 (CTCAE v 4.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 4.0
- Grade 3 (CTCAE v 4.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 4.0
- Grade 4 (CTCAE v 4.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 4.0
- Grade 5 (CTCAE v 4.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 4.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 4.0) | Grade 2 (CTCAE v 4.0) | Grade 3 (CTCAE v 4.0) | Grade 4 (CTCAE v 4.0) | Grade 5 (CTCAE v 4.0)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Participants
  Ear and labyrinth | 18 | 1 | 1 | 0 | 0 | 0
  Eye | 18 | 2 | 0 | 0 | 0 | 0
  Nausea | 6 | 10 | 3 | 1 | 0 | 0
  Vomiting | 13 | 6 | 0 | 1 | 0 | 0
  Abdominal pain | 13 | 4 | 1 | 2 | 0 | 0
  Other GI | 12 | 6 | 2 | 0 | 0 | 0
  Fever | 16 | 3 | 1 | 0 | 0 | 0
  Chills | 16 | 4 | 0 | 0 | 0 | 0
  Fatigue | 9 | 7 | 4 | 0 | 0 | 0
  General, NOS | 15 | 1 | 4 | 0 | 0 | 0
  Administrative site | 17 | 1 | 2 | 0 | 0 | 0
  Infections/infestations | 19 | 0 | 1 | 0 | 0 | 0
  Anorexia | 17 | 3 | 0 | 0 | 0 | 0
  Dehydration | 18 | 0 | 2 | 0 | 0 | 0
  Musculoskeletal/connective tissue | 17 | 2 | 1 | 0 | 0 | 0
  Peripheral Sensory neuropathy | 17 | 2 | 1 | 0 | 0 | 0
  Other nervous system | 17 | 3 | 0 | 0 | 0 | 0
  Psychiatric | 17 | 3 | 0 | 0 | 0 | 0
  Reproductive/breast | 19 | 1 | 0 | 0 | 0 | 0
  Respiratory/thoracic/mediastinal | 18 | 1 | 1 | 0 | 0 | 0
  Skin/subcutaneous | 16 | 4 | 0 | 0 | 0 | 0
  Leukopenia | 15 | 3 | 2 | 0 | 0 | 0
  Lymphopenia | 18 | 0 | 1 | 1 | 0 | 0
  Neutropenia | 15 | 5 | 0 | 0 | 0 | 0
  Thrombocytopenia | 13 | 6 | 1 | 0 | 0 | 0
  Anemia | 9 | 5 | 5 | 1 | 0 | 0
  Hyponatremia | 19 | 1 | 0 | 0 | 0 | 0
  Elevated Creatinine | 18 | 1 | 1 | 0 | 0 | 0
  Hyperglycemia | 19 | 1 | 0 | 0 | 0 | 0
  Hypomagnesemia | 18 | 2 | 0 | 0 | 0 | 0
  Hypoalbuminemia | 19 | 1 | 0 | 0 | 0 | 0
  Elevated alanine aminotransferase | 19 | 0 | 1 | 0 | 0 | 0
  Elevated alkaline phosphatase | 18 | 2 | 0 | 0 | 0 | 0
  Elevated aspartate aminotransferase | 18 | 1 | 1 | 0 | 0 | 0
  Elevated GGT | 19 | 0 | 1 | 0 | 0 | 0
  Elevated bilirubin | 19 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: The duration of time from start of treatment to time of death or the date of last contact, assessed up to 5 years
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (EGEN-001)
Number analyzed (Participants) | 20
months | 9.2 [5.7 to 16.3]

5. Secondary Outcome: Progression-free Survival
Description: The time from entry until disease progression, death, or date of last contact. Endpoints are progression or death. Patients who are not observed with an endpoint are censored.
Time Frame: The duration of time from start of treatment to time of progression or death, whichever occurs first, assessed up to 5 years
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (EGEN-001)
Number analyzed (Participants) | 20
months | 2.9 [2.0 to 6.3]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment
Arm/Group | Treatment (EGEN-001)
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (EGEN-001) (N=20)
Anemia (Blood and lymphatic system disorders) | 1
Colonic Obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3
Ileal Fistula (Gastrointestinal disorders) | 1
Death Nos (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Creatinine Increased (Investigations) | 3
White Blood Cell Decreased (Investigations) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (EGEN-001) (N=20)
Anemia (Blood and lymphatic system disorders) | 15
Palpitations (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Hearing Impaired (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Blurred Vision (Eye disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 8
Bloating (Gastrointestinal disorders) | 1
Anal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 9
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Pain (General disorders) | 6
Malaise (General disorders) | 3
Injection Site Reaction (General disorders) | 1
Infusion Site Extravasation (General disorders) | 2
Flu Like Symptoms (General disorders) | 1
Fatigue (General disorders) | 13
Fever (General disorders) | 4
Chills (General disorders) | 4
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 1
Weight Loss (Investigations) | 2
Platelet Count Decreased (Investigations) | 7
Lymphocyte Count Decreased (Investigations) | 2
Ggt Increased (Investigations) | 1
Creatinine Increased (Investigations) | 6
Neutrophil Count Decreased (Investigations) | 5
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 5
Aspartate Aminotransferase Increased (Investigations) | 3
Alkaline Phosphatase Increased (Investigations) | 4
Alanine Aminotransferase Increased (Investigations) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 4
Memory Impairment (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Depressed Level Of Consciousness (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 2
Bladder Spasm (Renal and urinary disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Nail Ridging (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1
Menopause (Reproductive system and breast disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hot Flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less